CLINICAL TRIAL: NCT06356129
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Comparing the Efficacy and Safety of Golcadomide Plus R-CHOP Chemotherapy vs Placebo Plus R-CHOP Chemotherapy in Participants With Previously Untreated High-risk Large B-cell Lymphoma (GOLSEEK-1)
Brief Title: Study to Compare the Effectiveness and Safety of Golcadomide Plus R-CHOP vs Placebo Plus R-CHOP in Participants With Previously Untreated High-risk Large B-cell Lymphoma
Acronym: GOLSEEK-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA073-1020; 2023-510178-15 (Registry Identifier: EU CT Number); U1111-1300-8493 (Registry Identifier: UTN)
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Large B-cell Lymphoma
Keywords: Lymphoma, Large B-Cell; Lymphoma; BMS-986369; CC-99282; DLBCL
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Golcadomide + R-CHOP (Rituximab, Doxorubicin, Vincristine, Cyclophosphamide, Prednisone) (Experimental)
  Interventions: Drug: Golcadomide; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Placebo + R-CHOP (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Golcadomide — Specified dose on specified days
  Other Names: BMS-986369; CC-99282
  Arms: Golcadomide + R-CHOP (Rituximab, Doxorubicin, Vincristine, Cyclophosphamide, Prednisone)
Drug: Placebo — Specified dose on specified days
  Arms: Placebo + R-CHOP
Drug: Rituximab — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days
Drug: Doxorubicin — Specified dose on specified days
Drug: Vincristine — Specified dose on specified days
Drug: Prednisone — Specified dose on specified days

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of golcadomide in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) chemotherapy vs placebo in combination with R-CHOP chemotherapy in participants with previously untreated high-risk large B-cell lymphoma (LBCL).

ELIGIBILITY:
Inclusion Criteria

- Histologically confirmed (per local evaluation) diagnosis of de novo, previously untreated large B-cell lymphoma (LBCL) according to 2022 world health organization (WHO) classification including:

i) Diffuse large B-cell lymphoma (DLBCL), not otherwise specified [including germinal center B-cell (GCB) and activated B-cell (ABC) types]

ii) High-grade B-cell lymphoma, with MYC and BCL2 rearrangements (HGBL-MYC/BCL2 double-hit lymphomas)

iii) High-grade B-cell lymphoma, not otherwise specified

iv) T-cell/histiocyte/rich large B-cell lymphoma (THRLBCL)

v) Epstein-Barr virus + DLBCL

* International Prognostic Index (IPI) score 1 or 2 with lactate dehydrogenase (LDH) > 1.3 x upper limit of normal (ULN) and/or bulky disease defined as single lesion of ≥ 7 cm OR IPI ≥ 3.
* Measurable disease defined by at least 1 fluorodeoxyglucose (FDG)-avid lesion for FDG-avid subtype and 1 bi-dimensionally measurable (> 1.5 cm in longest diameter) disease by computed tomography (CT) or magnetic resonance imaging (MRI), as defined by the Lugano classification.
* Must have Ann Arbor Stage II-IV disease.

Exclusion Criteria

* Any significant medical condition, active infection, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
* Any other subtype of lymphoma. Cases of primary mediastinal (thymic) large B-cell lymphoma (PMBCL), primary cutaneous DLBCL-leg type, Grade 3b FL, indolent lymphoma transformed to large B-cell lymphoma (LBCL), Anaplastic lymphoma kinase (ALK) positive large B-cell lymphoma, primary effusion lymphoma, and Burkitt lymphoma.
* Documented or suspected central nervous system (CNS) involvement by lymphoma.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2028-08-14 (Estimated); Study Completion 2029-11-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the Investigator | Up to approximately 67 months

SECONDARY OUTCOMES:
PFS assessed by the Investigator | Up to approximately 67 months
Overall survival (OS) | Up to approximately 67 months
Event-free survival (EFS) | Up to approximately 67 months
Complete Metabolic Response assessed by the Independent Response Adjudication Committee (IRAC) | Up to approximately 18 weeks
Minimal residual disease (MRD) negativity rate | Up to approximately 18 weeks
Progression-free survival (PFS) assessed by the IRAC | Up to approximately 47 months
Objective response (OR) assessed by the Investigator | Up to approximately 18 weeks
Complete metabolic response (CMR) assessed by the Investigator | Up to approximately 18 weeks
PFS24 assessed by the Investigator 24 months after randomization | Up to 24 months
Duration of response (DoR) | Up to approximately 67 months
Second progression-free survival (PFS2) assessed by the Investigator | Up to approximately 67 months
Relative dose intensity (%) | Up to 18 weeks
Time from randomization to meaningful improvement in primary domains of interest in the European Organization for Research and Treatment of Cancer - Quality of Life C30 (EORTC QLQ-C30) Questionnaire | Up to approximately 67 months
Time from randomization to meaningful improvement in primary domains of interest in the Functional Assessment of Cancer Treatment-Lymphoma (FACT-LymS) Questionnaire | Up to approximately 67 months
Mean change from baseline in the EORTC QLQ-C30 | Up to approximately 67 months
Mean change from baseline in the FACT-LymS | Up to approximately 67 months
Number of participants with Adverse Events (AEs) | Up to approximately 20 weeks
Number of participants with treatment-emergent adverse events (TEAEs) | Up to approximately 20 weeks
Number of participants with laboratory abnormalities | Up to approximately 20 weeks
Number of participants with vital sign abnormalities | Up to approximately 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (325):
- United States (46):
  - Local Institution - 0014, Mobile, Alabama
  - Local Institution - 0477, Anchorage, Alaska
  - Local Institution - 0452, Phoenix, Arizona
  - Local Institution - 0342, San Francisco, California
  - Local Institution - 0497, Fort Myers, Florida
  - Local Institution - 0287, Jacksonville, Florida
  - Local Institution - 0415, Margate, Florida
  - Local Institution - 0045, Miami Beach, Florida
  - Local Institution - 0012, Pensacola, Florida
  - Local Institution - 0502, St. Petersburg, Florida
  - Local Institution - 0414, Tampa, Florida
  - Local Institution - 0192, West Palm Beach, Florida
  - Local Institution - 0485, Weston, Florida
  - Local Institution - 0515, Atlanta, Georgia
  - Local Institution - 0303, Atlanta, Georgia
  - Local Institution - 0182, Chicago, Illinois
  - Local Institution - 0048, Skokie, Illinois
  - Local Institution - 0461, Waukee, Iowa
  - Local Institution - 0031, Westwood, Kansas
  - Local Institution - 0436, Edgewood, Kentucky
  - Local Institution - 0408, Baton Rouge, Louisiana
  - Local Institution - 0478, Ann Arbor, Michigan
  - Local Institution - 0067, Minneapolis, Minnesota
  - Local Institution - 0203, Rochester, Minnesota
  - Local Institution - 0437, Kansas City, Missouri
  - Local Institution - 0466, Reno, Nevada
  - Local Institution - 0498, East Brunswick, New Jersey
  - Local Institution - 0480, Hackensack, New Jersey
  - Local Institution - 0049, Morristown, New Jersey
  - Local Institution - 0175, New Brunswick, New Jersey
  - Local Institution - 0190, Buffalo, New York
  - Local Institution - 0451, East Syracuse, New York
  - Local Institution - 0484, New York, New York
  - Local Institution - 0369, New York, New York
  - Local Institution - 0176, New York, New York
  - Local Institution - 0174, Chapel Hill, North Carolina
  - Local Institution - 0066, Massillon, Ohio
  - Local Institution - 0450, Tulsa, Oklahoma
  - Local Institution - 0179, Portland, Oregon
  - Local Institution - 0009, Pittsburgh, Pennsylvania
  - Local Institution - 0419, York, Pennsylvania
  - Local Institution - 0435, Fort Sam Houston, Texas
  - Local Institution - 0516, Houston, Texas
  - Local Institution - 0046, Houston, Texas
  - Local Institution - 0424, Houston, Texas
  - Local Institution - 0293, Richmond, Virginia
- Argentina (6):
  - Local Institution - 0113, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0421, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0112, Buenos Aires
  - Local Institution - 0119, Buenos Aires
  - Local Institution - 0136, Buenos Aires
  - Local Institution - 0111, Córdoba
- Australia (10):
  - Local Institution - 0357, Gosford, New South Wales
  - Local Institution - 0361, Sydney, New South Wales
  - Local Institution - 0358, Westmead, New South Wales
  - Local Institution - 0363, Tiwi, Northern Territory
  - Local Institution - 0356, Birtinya, Queensland
  - Local Institution - 0360, Southport, Queensland
  - Local Institution - 0365, Frankston, Victoria
  - Local Institution - 0362, Heidelberg, Victoria
  - Local Institution - 0359, St Albans, Victoria
  - Local Institution - 0364, Warrnambool, Victoria
- Austria (3):
  - Local Institution - 0385, Wels, Upper Austria
  - Local Institution - 0387, Linz
  - Local Institution - 0386, Vienna
- Brazil (19):
  - Local Institution - 0255, Fortaleza, Ceará
  - Local Institution - 0297, Lago Sul, Federal District
  - Local Institution - 0256, Goiânia, Goiás
  - Local Institution - 0302, Curitiba, Paraná
  - Local Institution - 0296, Niterói, Rio de Janeiro
  - Local Institution - 0304, Natal, Rio Grande do Norte
  - Local Institution - 0253, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0246, Chapecó, Santa Catarina
  - Local Institution - 0247, Joinville, Santa Catarina
  - Local Institution - 0250, Barretos, São Paulo
  - Local Institution - 0249, Jaú, São Paulo
  - Local Institution - 0301, São José do Rio Preto, São Paulo
  - Local Institution - 0248, São Paulo, São Paulo
  - Local Institution - 0316, São Paulo, São Paulo
  - Local Institution - 0298, Rio de Janeiro
  - Local Institution - 0294, São Paulo
  - Local Institution - 0252, São Paulo
  - Local Institution - 0317, São Paulo
  - Local Institution - 0251, São Paulo
- Bulgaria (3):
  - Local Institution - 0393, Plovdiv
  - Local Institution - 0392, Sofia
  - Local Institution - 0394, Sofia
- Canada (4):
  - Local Institution - 0091, Victoria, British Columbia
  - Local Institution - 0153, Montreal, Quebec
  - Local Institution - 0073, Montreal, Quebec
  - Local Institution - 0004, Sherbrooke, Quebec
- Chile (6):
  - Local Institution - 0164, Viña del Mar, Región de Valparaíso
  - Local Institution - 0106, Santiago, Santiago Metropolitan
  - Local Institution - 0107, Santiago, Santiago Metropolitan
  - Local Institution - 0108, Santiago, Santiago Metropolitan
  - Local Institution - 0110, Santiago, Santiago Metropolitan
  - Local Institution - 0459, Santiago, Santiago Metropolitan
- China (30):
  - Local Institution - 0195, Beijing, Beijing Municipality
  - Local Institution - 0236, Chongqing, Chongqing Municipality
  - Local Institution - 0196, Chongqing, Chongqing Municipality
  - Local Institution - 0274, Fuzhou, Fujian
  - Local Institution - 0157, Xiamen, Fujian
  - Local Institution - 0133, Guangzhou, Guangdong
  - Local Institution - 0240, Guangzhou, Guangdong
  - Local Institution - 0338, Nanning, Guangxi
  - Local Institution - 0239, Harbin, Heilongjiang
  - Local Institution - 0238, Zhengzhou, Henan
  - Local Institution - 0346, Wuhan, Hubei
  - Local Institution - 0214, Wuhan, Hubei
  - Local Institution - 0275, Changsha, Hunan
  - Local Institution - 0156, Suzhou, Jiangsu
  - Local Institution - 0237, Nanchang, Jiangxi
  - Local Institution - 0241, Nanchang, Jiangxi
  - Local Institution - 0291, Changchun, Jilin
  - Local Institution - 0334, Shenyang, Liaoning
  - Local Institution - 0169, Shenyang, Liaoning
  - Local Institution - 0242, Jinan, Shandong
  - Local Institution - 0344, Jinan, Shandong
  - Local Institution - 0132, Shanghai, Shanghai Municipality
  - Local Institution - 0339, Shanghai, Shanghai Municipality
  - Local Institution - 0234, Taiyuan, Shanxi
  - Local Institution - 0141, Chengdu, Sichuan
  - Local Institution - 0470, Tianjin, Tianjin Municipality
  - Local Institution - 0467, Ürümqi, Xinjiang
  - Local Institution - 0197, Hangzhou, Zhejiang
  - Local Institution - 0483, Hangzhou, Zhejiang
  - Local Institution - 0457, Wenzhou, Zhejiang
- Colombia (2):
  - Local Institution - 0129, Bogotá, Bogota D.C.
  - Local Institution - 0130, Bogota, Cundinamarca
- Czechia (6):
  - Local Institution - 0105, Brno, Brno-město
  - Local Institution - 0104, Hradec Králové, Hradec Králové
  - Local Institution - 0102, Olomouc, Olomoucký kraj
  - Local Institution - 0120, Pilsen, Plzeň Region
  - Local Institution - 0103, Prague, Praha 10
  - Local Institution - 0243, Prague
- Denmark (2):
  - Local Institution - 0285, Aarhus, Central Jutland
  - Local Institution - 0284, Odense, Region Syddanmark
- Finland (4):
  - Local Institution - 0281, Oulu, North Ostrobothnia
  - Local Institution - 0283, Kuopio, Northern Savonia
  - Local Institution - 0282, Turku, Southwest Finland
  - Local Institution - 0280, Helsinki
- France (24):
  - Local Institution - 0083, Nice, Alpes-Maritimes
  - Local Institution - 0084, Strasbourg, Alsace
  - Local Institution - 0090, Bordeaux, Aquitaine
  - Local Institution - 0324, Pessac, Aquitaine
  - Local Institution - 0087, Marseille, Bouches-du-Rhône
  - Local Institution - 0292, Dijon, Côte-d'Or
  - Local Institution - 0486, Besançon, Doubs
  - Local Institution - 0332, Brest, Finistère
  - Local Institution - 0202, Lille, Hauts-de-France
  - Local Institution - 0335, Saint-Cloud, Hauts-de-Seine
  - Local Institution - 0079, Tours, Indre-et-Loire
  - Local Institution - 0223, La Tronche, Isère
  - Local Institution - 0323, Saint-Pierre, La Réunion
  - Local Institution - 0074, Montpellier, Languedoc-Roussillon
  - Local Institution - 0081, Lille, Nord
  - Local Institution - 0325, Nantes, Pays de la Loire Region
  - Local Institution - 0321, Saint Priest En Jarez, Pays de la Loire Region
  - Local Institution - 0089, Pierre-Bénite, Rhône
  - Local Institution - 0200, Créteil, Val-de-Marne
  - Local Institution - 0076, Villejuif, Val-de-Marne
  - Local Institution - 0306, Poitiers, Vienne
  - Local Institution - 0244, Bayonne
  - Local Institution - 0315, Caen
  - Local Institution - 0077, Paris
- Germany (13):
  - Local Institution - 0511, Ulm, Baden-Wurttemberg
  - Local Institution - 0383, Augsburg, Bavaria
  - Local Institution - 0512, Bayreuth, Bavaria
  - Local Institution - 0505, Erlangen, Bavaria
  - Local Institution - 0507, Langen, Hesse
  - Local Institution - 0513, Hanover, Lower Saxony
  - Local Institution - 0384, Koblenz, Rhineland-Palatinate
  - Local Institution - 0504, Halle, Saxony-Anhalt
  - Local Institution - 0506, Lübeck, Schleswig-Holstein
  - Local Institution - 0508, Berlin
  - Local Institution - 0503, Cottbus
  - Local Institution - 0510, Dresden
  - Local Institution - 0370, Essen
- Greece (5):
  - Local Institution - 0398, Alexandroupoli, Anatolikí Makedonía Kai Thráki
  - Local Institution - 0399, Athens, Attikí
  - Local Institution - 0396, Athens, Attikí
  - Local Institution - 0397, Chaïdári, Attikí
  - Local Institution - 0395, Ioannina, Ípeiros
- Hungary (6):
  - Local Institution - 0266, Debrecen, Hajdú-Bihar
  - Local Institution - 0162, Kaposvár, Somogy County
  - Local Institution - 0353, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Local Institution - 0161, Szombathely, Vas County
  - Local Institution - 0163, Budapest
  - Local Institution - 0160, Budapest
- India (7):
  - Local Institution - 0411, Belagavi, Karnataka
  - Local Institution - 0430, Kochi, Kerala
  - Local Institution - 0154, Mumbai, Maharashtra
  - Local Institution - 0433, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0469, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0413, Howrah, West Bengal
  - Local Institution - 0410, New Town, West Bengal
- Italy (4):
  - Local Institution - 0495, Ravenna, Emilia-Romagna
  - Local Institution - 0493, Rome, Lazio
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO, Palermo, Sicily
  - Local Institution - 0496, Novara
- Japan (29):
  - Local Institution - 0371, Nagoya, Aichi-ken
  - Local Institution - 0168, Kashiwa, Chiba
  - Local Institution - 0475, Eiheiji-cho,Yoshida-gun, Fukui
  - Local Institution - 0271, Ōgaki, Gifu
  - Local Institution - 0368, Sapporo, Hokkaido
  - Local Institution - 0327, Sapporo, Hokkaido
  - Local Institution - 0273, Amagasaki, Hyōgo
  - Local Institution - 0328, Himeji, Hyōgo
  - Local Institution - 0270, Kanazawa, Ishikawa-ken
  - Local Institution - 0343, Morioka, Iwate
  - Local Institution - 0170, Isehara, Kanagawa
  - Local Institution - 0333, Yokohama, Kanagawa
  - Local Institution - 0320, Sendai, Miyagi
  - Local Institution - 0166, Sakai, Osaka
  - Local Institution - 0269, Hidaka, Saitama
  - Local Institution - 0288, Nagaizumi-cho,Sunto-gun, Shizuoka
  - Local Institution - 0350, Bunkyo-ku, Tokyo
  - Local Institution - 0268, Itabashiku, Tokyo
  - Local Institution - 0331, Chūō, Yamanashi
  - Local Institution - 0348, Fukuoka
  - Local Institution - 0319, Fukuoka
  - Local Institution - 0313, Fukuoka
  - Local Institution - 0272, Hiroshima
  - Local Institution - 0171, Kumamoto
  - Local Institution - 0215, Kyoto
  - Local Institution - 0329, Okayama
  - Local Institution - 0322, Osaka
  - Local Institution - 0347, Osaka
  - Local Institution - 0167, Yamagata
- Malaysia (4):
  - Local Institution - 0453, Lembah Pantai, Kuala Lumpur
  - Local Institution - 0432, George Town, Pulau Pinang
  - Local Institution - 0431, Kuching, Sarawak
  - Local Institution - 0449, Ampang, Selangor
- Mexico (8):
  - Local Institution - 0122, Mexico City, DIF
  - Local Institution - 0121, Mexico City, DIF
  - Local Institution - 0128, Mexico City, Mexico City
  - Local Institution - 0126, Mexico City, Mexico City
  - Local Institution - 0127, Morelia, Michoacán
  - Local Institution - 0139, Monterrey, Nuevo León
  - Local Institution - 0125, Oaxaca City, Oaxaca
  - Local Institution - 0124, Puebla City
- Netherlands (2):
  - Local Institution - 0500, Leiden, South Holland
  - Local Institution - 0499, Groningen
- New Zealand (3):
  - Local Institution - 0367, Dunedin, Otago
  - Local Institution - 0366, Hamilton, Waikato Region
  - Local Institution - 0462, Auckland
- Local Institution - 0391, Oslo, Norway
- Poland (6):
  - Local Institution - 0388, Skórzewo, Greater Poland Voivodeship
  - Local Institution - 0336, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0201, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0337, Lublin, Lublin Voivodeship
  - Local Institution - 0443, Warsaw, Masovian Voivodeship
  - Local Institution - 0330, Katowice, Silesian Voivodeship
- Portugal (2):
  - Local Institution - 0286, Lisbon
  - Local Institution - 0098, Porto
- Local Institution - 0372, San Juan, Puerto Rico
- Romania (10):
  - Local Institution - 0381, Bucharest, București
  - Local Institution - 0417, Tg.Mures, Mureș County
  - Local Institution - 0380, Brasov
  - Local Institution - 0374, Bucharest
  - Local Institution - 0377, Bucharest
  - Local Institution - 0382, Bucharest
  - Local Institution - 0378, Bucharest
  - Local Institution - 0423, Cluj-Napoca
  - Local Institution - 0379, Iași
  - Local Institution - 0376, Sibiu
- Saudi Arabia (4):
  - Local Institution - 0439, Dammam, Eastern Province
  - Local Institution - 0445, Riyadh, Riyadh Region
  - Local Institution - 0438, Jeddah
  - Local Institution - 0416, Riyadh
- Local Institution - 0427, Singapore, Central Singapore, Singapore
- Local Institution - 0204, Bratislava, Slovakia
- South Korea (13):
  - Local Institution - 0149, Goyang-si, Kyǒnggi-do
  - Local Institution - 0456, Seongnam, Kyǒnggi-do
  - Local Institution - 0233, Suwon, Kyǒnggi-do
  - Local Institution - 0115, Busan, Pusan-Kwangyǒkshi
  - Local Institution - 0114, Busan, Pusan-Kwangyǒkshi
  - Local Institution - 0131, Busan, Pusan-Kwangyǒkshi
  - Local Institution - 0143, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0069, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0100, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0068, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0070, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0441, Deagu, Taegu-Kwangyǒkshi
  - Local Institution - 0118, Seoul
- Spain (15):
  - Local Institution - 0412, A Coruña, A Coruña [La Coruña]
  - Local Institution - 0491, Badalona, Barcelona [Barcelona]
  - Local Institution - 0071, L'Hospitalet Del Llobregat, Barcelona [Barcelona]
  - Local Institution - 0389, Barakaldo, Bizkaia
  - Local Institution - 0172, Santa Cruz de Tenerife, Canary Islands
  - Local Institution - 0314, Donostia / San Sebastian, Gipuzkoa
  - Local Institution - 0096, Majadahonda, Madrid, Comunidad de
  - Local Institution - 0409, El Palmar, Murcia, Murcia, Región de
  - Local Institution - 0092, Málaga, Málaga
  - Local Institution - 0095, Cáceres
  - Local Institution - 0072, Madrid
  - Local Institution - 0490, Madrid
  - Local Institution - 0488, Madrid
  - Local Institution - 0093, Salamanca
  - Local Institution - 0489, Seville
- Sweden (4):
  - Local Institution - 0279, Lund, Skåne Län [se-12]
  - Local Institution - 0487, Solna, Stockholms Län [se-01]
  - Local Institution - 0277, Uppsala, Uppsala Län [se-03]
  - Local Institution - 0278, Linköping, Östergötlands Län [se-05]
- Taiwan (9):
  - Local Institution - 0142, Chiayi City, Chiayi
  - Local Institution - 0146, Tainan, Tainan
  - Local Institution - 0159, Kaohsiung City
  - Local Institution - 0135, Taichung
  - Local Institution - 0145, Taichung
  - Local Institution - 0134, Taipei
  - Local Institution - 0514, Taipei
  - Local Institution - 0147, Taipei
  - Local Institution - 0158, Taoyuan District
- Thailand (4):
  - Local Institution - 0434, Bangkok, Bangkok
  - Ramathibodi Hospital, Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital, Bangkok, Bangkok
  - Local Institution - 0428, Chiang Mai
- Turkey (Türkiye) (8):
  - Local Institution - 0400, Ankara
  - Local Institution - 0405, Ankara
  - Local Institution - 0422, Ankara
  - Local Institution - 0401, Ankara
  - Local Institution - 0406, Izmir
  - Local Institution - 0403, Mersin
  - Local Institution - 0407, Samsun
  - Local Institution - 0402, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06356129.html